CLINICAL TRIAL: NCT01255176
Title: Evaluation of the Effects of Physical Therapy Method of Restoring Cardiac Thoracic Abdominal Infants
Brief Title: Rebalancing Thoraco Abdominal Heart Disease in Infants (RTAC)
Acronym: RTAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Camila Isabel Santos Schivinski, Dr., University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEMFRTALC2010
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2010-12

CONDITIONS: Infants With Heart Disease; Respiratory Therapy; Techniques
Keywords: Infant; Physical Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo group (No Intervention): not receive physical therapy intervention, there will only support the achievement of a handbook on the abdomen of the baby.
- control group (No Intervention): not receive any type of intervention, and infants remain at rest
- Thoracoabdominal rebalancing (Experimental): infants who receive physical therapy through the application of the handlings of the RTA.
  Interventions: Procedure: Thoracoabdominal rebalancing

INTERVENTIONS:
Procedure: Thoracoabdominal rebalancing — In this group the infants received four handlings thoracoabdominal rebalancing, in order: 1) 5min support thoracoabdominal, in which the therapist leaned one hand on the lower chest and upper abdomen of the newborn, with some of its fingers on the ribs, pulling them gently down and keeping them in that position during inspiration, 2) more than 5 minutes of abdominal support, carried by hand in the lower abdomen of the newborn, applying light pressure during inspiration enough to be beaten by the diaphragm of the newborn and not to increase the use of accessory muscles of inspiration, 3) 5min support ileo-costal, by a slight manual pressure of the physiotherapist on the lateral chest and abdomen of the newborn, maintained throughout inspiration and 4) finally ran up 5min ginga thoracic maneuver slight manual pressure on the lower chest of newborns, directing the costal movement during expiration, now an then the other hemithorax.
  Arms: Thoracoabdominal rebalancing

SUMMARY:
It gave a clinical trial which will be included in the 60 infants, aged up to 24 months, diagnosed with congenital's population will be divided by simple randomization into three groups: 20 infants in the intervention group, 20 infants in the control group, not receive the RTA technique and another 20 infants in a placebo group, we just get the support manual therapist for 5 minutes. Initially the data will be collected cardio heart rate, respiratory rate and oxygen saturation. Then the researcher will apply three specific rating scales, based on clinical presentation and behavior of infants. Hypothesis: The RTA improves cardiorespiratory parameters and reduces signs of discomfort and pain of infants with congenital heart acyanogenic.

ELIGIBILITY:
Inclusion Criteria:

* Newborns admitted to the nursery without ventilatory support or oxygen therapy, and whose parents agree with the child's participation in the study. Will be excluded newborns who have some problems during any of the study procedures and those whose condition will change after the intervention, with shift in ventilatory support or oxygen therapy.

Exclusion Criteria:

* In case of inability to collect some of the parameters evaluated at the appropriate time, the RN also will no longer part of the sample, as well as those who show no contraindication to therapy.

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in cardiorespiratory parameters | 15 minutes after the end of the intervention
Pain Scales (NIPS, PIPP, NFCS) | Immediately after intervention and 15 minutes after the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Camila Schivinski, Doctor, Principal Investigator — Professor of Universidade do Estado de Santa Catarina
Locations (1):
- Joana de Gusmão Children's Hospital, Florianópolis, Santa Catarina, Brazil